CLINICAL TRIAL: NCT03184545
Title: A Prospective Randomized Study Comparing the Outcome of Electrical Stimulation of Vastus Medialis Obliquus Muscle and Physical Therapy Vs Only Physical Therapy but No Electrical Stimulation in Patients with Patellofemoral Pain Syndrome
Brief Title: Comparing the Outcome of Electrical Stimulation and Physical Therapy in Patellofemoral Pain Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Leon Popovitz, Orthopaedic Surgeon, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-726
Record Dates: First submitted 2017-06-04; First posted 2017-06-12 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: anterior knee pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: It's a phase III study. A randomized, observer blinded, single center study. Patients will be divided in two groups based on randomization. One group will receive electrical muscle stimulation and Physical therapy and other group will receive only physical therapy. Electrical muscle stimulation device is The Flex MT Plus (Electrostim Medical Services Inc. Tampa, FL) is a neuromuscular stimulator. It is approved by the Food and Drug Administration (FDA). Assessment and follow up will be performed before start of treatment, at 3 weeks, 6 weeks, 12 weeks, 6 months and 12 months post-start of treatment . Assessment will be done at each visit based on Kujala patellofemoral score, pain visual analog scale (VAS) during activities of daily life and isometric strength measurement.
Who Masked: Outcomes Assessor
Masking Description: The examiner who will be evaluating and assessing the outcome scores on each visit will be blinded to the patient's group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EMS and PT (Experimental): Group 1: Electrical Muscle stimulation (EMS) and Physical therapy (PT).
  Interventions: Device: EMS; Other: Physical therapy
- Only PT (Active Comparator): Group 2: Only Physical therapy (PT).
  Interventions: Other: Physical therapy

INTERVENTIONS:
Device: EMS — The EMS device Flex MT Plus (Electrostim Medical Services Inc. Tampa, FL) is a neuromuscular stimulator. It is approved by the FDA. The Electrical muscle stimulation (EMS) applied to vastus medialis obliquus (VMO) muscle for 20 minutes, 3 times daily and it would be 5 times a week for 12 weeks at 40 Hz. The pulse duration will be 0.26ms, at 5 seconds on and 10 seconds off.
  Arms: EMS and PT
Other: Physical therapy — Standard physical therapy exercises

SUMMARY:
The purpose of study is to evaluate the efficacy of the electrical muscle stimulation (EMS) device in patients with patellofemoral pain known as anterior knee pain. Usual treatment for it is physical therapy (PT). We want to evaluate and see if adding the electrical muscle stimulation will fasten the recovery and improved outcome in patellofemoral pain syndrome. Half of participants will receive EMS and PT while other half will receive PT only.

DETAILED DESCRIPTION:
The patellofemoral pain syndrome also known as anterior knee pain is a common entity in young athletic population. In patellofemoral knee syndrome, one of the theory is that the vastus medialis obliquus muscle is weak. To strengthen the muscle, physical therapy exercises are commonly used. This study evaluates addition of the electrical muscle stimulation device.The electrical muscle stimulation device "Flex MT Plus" (Electrostim Medical Services Inc. Tampa, FL) is a FDA approved device and has been used in knee for other conditions like treating for weakness associated with knee injuries or after knee surgeries. It has shown to improve the outcomes in above mentioned conditions. Its efficacy has been tested in patellofemoral pain syndrome but in smaller sample size. We intend to test it in larger sample size patient population.

Bily et al (2008) (reference #1) published their results on patellofemoral pain syndrome comparing EMS +PT to PT only and found that overall significant improvement in outcome score in all patients but when compared between the groups there was no difference. But there sample size was 19 patients in each group. Small sample size was one of the limitation of their study. We intend to collect 46 patients in each group to find significant difference based on power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral/unilateral anterior knee pain for more than 3 moths
* Age of patient 18 to 40 years
* At least 3 of the 4 following criteria present: pain associated with prolonged sitting with knees bend, pain with going downstairs, kneeling and squatting or sports activities
* No h/o injury
* No h/o surgery to the knee

Exclusion Criteria:

* H/o patellar dislocation or subluxation
* Associated bursitis, tendinitis in periarticular area
* Ligamentous problems
* Intra-articular pathology
* Pregnancy (patient reported pregnancy, in case of doubt patient will be referred to their OBG/GYN physician to exclude the pregnancy)
* H/o knee surgery
* Oral or intraarticular administration of steroid medication with in last 3 months
* Patients with implanted devices like pacemaker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Kujala patellofemoral score. | 2 years. Total duration of study is two years. But each patient will be followed for total 12 months after enrollment. If any patient enrolled at 1 year mark after start of study , he will be followed for one year. So total duration of study is 2 years.
  Assessment will be done at each visit (pre-treatment, post-start treatment 3 weeks,, 6 weeks, 12 weeks, 6 months and 12 months) based on Kujala patellofemoral score. The Kujala score assesses following points: Limp, support, walking, stairs, squatting,running, jumping, prolong sitting with knee flexed,pain,swelling,abnormal painful kneecap movements, atrophy of thigh and flexion deficiency. Repeated measures linear regression models will be used to compare the two treatment arms with respect to knee function, pain score, and muscle strength from baseline to 12 months.
  Total duration of study is two years. We intend finish enrolling 92 patients by the end of one year after start of study. But each patient will be followed for total 12 months period. If any patient enrolled at 1 year mark after start of study , he will be followed for one year.
Visual analog pain scale (VAS) pain scale during activities of life | 2 years
  VAS scale of 1-10 will be used to evaluate knee pain. 1 being mild and 10 being worst.
Isometric strength measurement of knee | 2 years
  Isometric strength will be measured using dynamo-meter.

SECONDARY OUTCOMES:
Secondary outcome measure would be how many return to sports activity. | 2 years
  Secondary outcome assessment will be to see how many in EMS+PT group and how many in PT group returned to their previous activity level of sports without any pain after completion of treatment.
At what point of time they returned to their sports activity | 2 years
  It will be also noted and compared between the groups at what time period after the start of treatment they returned to their regular sports activities. We hypothesize that EMS group might return early.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Popovitz, MD, Principal Investigator — Northwell Health
Locations (1):
- New York Bone and Joint Specialists, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No patient data will be shared.

REFERENCES:
- [Background] Bily W, Trimmel L, Modlin M, Kaider A, Kern H. Training program and additional electric muscle stimulation for patellofemoral pain syndrome: a pilot study. Arch Phys Med Rehabil. 2008 Jul;89(7):1230-6. doi: 10.1016/j.apmr.2007.10.048. PMID 18586125
- [Background] Callaghan MJ, Oldham JA, Winstanley J. A comparison of two types of electrical stimulation of the quadriceps in the treatment of patellofemoral pain syndrome. A pilot study. Clin Rehabil. 2001 Dec;15(6):637-46. doi: 10.1191/0269215501cr457oa. PMID 11777094
- [Background] Avramidis K, Strike PW, Taylor PN, Swain ID. Effectiveness of electric stimulation of the vastus medialis muscle in the rehabilitation of patients after total knee arthroplasty. Arch Phys Med Rehabil. 2003 Dec;84(12):1850-3. doi: 10.1016/s0003-9993(03)00429-5. PMID 14669193
- [Background] Callaghan MJ, Oldham JA. Electric muscle stimulation of the quadriceps in the treatment of patellofemoral pain. Arch Phys Med Rehabil. 2004 Jun;85(6):956-62. doi: 10.1016/j.apmr.2003.07.021. PMID 15179650
- [Background] Kuru T, Yaliman A, Dereli EE. Comparison of efficiency of Kinesio(R) taping and electrical stimulation in patients with patellofemoral pain syndrome. Acta Orthop Traumatol Turc. 2012;46(5):385-92. doi: 10.3944/aott.2012.2682. PMID 23268824
- [Background] Garcia FR, Azevedo FM, Alves N, Carvalho AC, Padovani CR, Negrao Filho RF. Effects of electrical stimulation of vastus medialis obliquus muscle in patients with patellofemoral pain syndrome: an electromyographic analysis. Rev Bras Fisioter. 2010 Nov-Dec;14(6):477-82. English, Portuguese. PMID 21340241
- [Background] Witvrouw E, Werner S, Mikkelsen C, Van Tiggelen D, Vanden Berghe L, Cerulli G. Clinical classification of patellofemoral pain syndrome: guidelines for non-operative treatment. Knee Surg Sports Traumatol Arthrosc. 2005 Mar;13(2):122-30. doi: 10.1007/s00167-004-0577-6. Epub 2005 Feb 10. PMID 15703965
- [Background] Avraham F, Aviv S, Ya'akobi P, Faran H, Fisher Z, Goldman Y, Neeman G, Carmeli E. The efficacy of treatment of different intervention programs for patellofemoral pain syndrome--a single blinded randomized clinical trial. Pilot study. ScientificWorldJournal. 2007 Aug 24;7:1256-62. doi: 10.1100/tsw.2007.167. PMID 17721640
- [Background] Chiu JK, Wong YM, Yung PS, Ng GY. The effects of quadriceps strengthening on pain, function, and patellofemoral joint contact area in persons with patellofemoral pain. Am J Phys Med Rehabil. 2012 Feb;91(2):98-106. doi: 10.1097/PHM.0b013e318228c505. PMID 22248804
- [Background] Rixe JA, Glick JE, Brady J, Olympia RP. A review of the management of patellofemoral pain syndrome. Phys Sportsmed. 2013 Sep;41(3):19-28. doi: 10.3810/psm.2013.09.2023. PMID 24113699
- [Background] Peng HT, Song CY. Predictors of treatment response to strengthening and stretching exercises for patellofemoral pain: An examination of patellar alignment. Knee. 2015 Dec;22(6):494-8. doi: 10.1016/j.knee.2014.10.012. Epub 2014 Nov 10. PMID 26254693
- [Background] Van Der Heijden RA, Lankhorst NE, Van Linschoten R, Bierma-Zeinstra SM, Van Middelkoop M. Exercise for treating patellofemoral pain syndrome: an abridged version of Cochrane systematic review. Eur J Phys Rehabil Med. 2016 Feb;52(1):110-33. Epub 2015 Jul 9. PMID 26158920
- [Background] Selhorst M, Rice W, Degenhart T, Jackowski M, Tatman M. Evaluation of a treatment algorithm for patients with patellofemoral pain syndrome: a pilot study. Int J Sports Phys Ther. 2015 Apr;10(2):178-88. PMID 25883866
- [Background] Alba-Martin P, Gallego-Izquierdo T, Plaza-Manzano G, Romero-Franco N, Nunez-Nagy S, Pecos-Martin D. Effectiveness of therapeutic physical exercise in the treatment of patellofemoral pain syndrome: a systematic review. J Phys Ther Sci. 2015 Jul;27(7):2387-90. doi: 10.1589/jpts.27.2387. Epub 2015 Jul 22. PMID 26311988
- [Background] Giles LS, Webster KE, McClelland JA, Cook J. Atrophy of the Quadriceps Is Not Isolated to the Vastus Medialis Oblique in Individuals With Patellofemoral Pain. J Orthop Sports Phys Ther. 2015 Aug;45(8):613-9. doi: 10.2519/jospt.2015.5852. Epub 2015 Jun 25. PMID 26110547
- [Background] Giles LS, Webster KE, McClelland JA, Cook J. Does quadriceps atrophy exist in individuals with patellofemoral pain? A systematic literature review with meta-analysis. J Orthop Sports Phys Ther. 2013 Nov;43(11):766-76. doi: 10.2519/jospt.2013.4833. Epub 2013 Sep 9. PMID 24175596
- [Background] Servodio Iammarrone C, Cadossi M, Sambri A, Grosso E, Corrado B, Servodio Iammarrone F. Is there a role of pulsed electromagnetic fields in management of patellofemoral pain syndrome? Randomized controlled study at one year follow-up. Bioelectromagnetics. 2016 Feb;37(2):81-8. doi: 10.1002/bem.21953. Epub 2016 Jan 12. PMID 26756278
- [Background] Ramazzina I, Pogliacomi F, Bertuletti S, Costantino C. Long term effect of selective muscle strengthening in athletes with patellofemoral pain syndrome. Acta Biomed. 2016 Apr 15;87 Suppl 1:60-8. PMID 27104322
- [Background] Chang WD, Huang WS, Lai PT. Muscle Activation of Vastus Medialis Oblique and Vastus Lateralis in Sling-Based Exercises in Patients with Patellofemoral Pain Syndrome: A Cross-Over Study. Evid Based Complement Alternat Med. 2015;2015:740315. doi: 10.1155/2015/740315. Epub 2015 Oct 4. PMID 26504480
- [Background] Fagan V, Delahunt E. Patellofemoral pain syndrome: a review on the associated neuromuscular deficits and current treatment options. Br J Sports Med. 2008 Oct;42(10):789-95. doi: 10.1136/bjsm.2008.046623. Epub 2008 Apr 18. PMID 18424487
- [Background] Crossley KM, Callaghan MJ, van Linschoten R. Patellofemoral pain. BMJ. 2015 Nov 4;351:h3939. doi: 10.1136/bmj.h3939. No abstract available. PMID 26537829
- [Background] Hott A, Liavaag S, Juel NG, Brox JI. Study protocol: a randomised controlled trial comparing the long term effects of isolated hip strengthening, quadriceps-based training and free physical activity for patellofemoral pain syndrome (anterior knee pain). BMC Musculoskelet Disord. 2015 Feb 25;16:40. doi: 10.1186/s12891-015-0493-6. PMID 25879452